CLINICAL TRIAL: NCT04759222
Title: Microvascular Reactivity as a Predictor of Major Adverse Events in Patients With On-pump Cardiac Surgery: A Prospective Observational Study
Brief Title: Microvascular Reactivity in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeon-Jeong Lee, Professor, Pusan National University Hospital
Other Study IDs: 1702-003-051
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: vascular occlusion test — The VOT was performed five times in each patient, before the induction of general anesthesia (baseline, T0), 30 min after the induction of general anesthesia (T1), 30 min after applying CPB (T2), 10 min after injection of protamine (T3), and after sternal closure (T4). Before induction of anesthesia, an NIRS sensor was placed on the thenar eminence and an automated tourniquet was placed around the upper arm. The arterial catheter was placed in the contralateral radial artery and the baseline blood pressure was measured. When the baseline tissue oxygen saturation (StO2) was stabilized, the automatic tourniquet was inflated to 50 mmHg over the patient's baseline systolic blood pressure and maintained for 5 min. After the 5-min ischemic period, the tourniquet rapidly deflated to 0 mmHg. StO2 data were continuously recorded during the VOT procedure.

SUMMARY:
Microcirculatory disturbance occurs most seriously during cardiopulmonary bypass (CPB) in cardiac surgery. If microvascular reactivity compensates for microcirculatory disturbance during CPB, tissue hypoxemia may be minimized. On the other hand, tissue hypoxemia may develop and lead to poor clinical outcomes. The primary aim of this study was to assess whether microvascular reactivity during CPB can predict major adverse events (MAE) within 30 days after cardiac surgery.

This prospective, observational, single-center study was conducted on 115 patients who underwent elective on-pump cardiac surgery. The vascular occlusion test (VOT) with near-infrared spectroscopy was performed five times for each patient, before the induction of general anesthesia (baseline, T0), 30 min after the induction of general anesthesia (T1), 30 min after applying CPB (T2), 10 min after injection of protamine (T3), and after sternal closure (T4). Sequential Organ Failure Assessment (SOFA) and Acute Physiologic and Chronic Health Evaluation (APACHE) II scores and the length of ventilator care, intensive care unit stay, and hospital stay were recorded. Postoperative MAE within 30 days after surgery was also recorded.

DETAILED DESCRIPTION:
The VOT was performed five times in each patient, before the induction of general anesthesia (baseline, T0), 30 min after the induction of general anesthesia (T1), 30 min after applying CPB (T2), 10 min after injection of protamine (T3), and after sternal closure (T4). Before induction of anesthesia, an NIRS sensor (INVOS® 5100C Cerebral/Somatic Oximeter; Medtronic, Minneapolis, MN, USA) was placed on the thenar eminence and an automated tourniquet (A.T.S® 3000 Automatic Tourniquet System; Zimmer Inc., Warsaw, IL, USA) was placed around the upper arm. The arterial catheter was placed in the contralateral radial artery and the baseline blood pressure was measured. When the baseline tissue oxygen saturation (StO2) was stabilized, the automatic tourniquet was inflated to 50 mmHg over the patient's baseline systolic blood pressure and maintained for 5 min. After the 5-min ischemic period, the tourniquet rapidly deflated to 0 mmHg. StO2 data were continuously recorded during the VOT procedure. Baseline StO2, minimum StO2 during the 5-min inflation of the tourniquet, and maximum StO2 during deflation of the tourniquet were obtained. The occlusion slope and recovery slope were calculated based on the measured StO2 data. The occlusion slope, which is related to oxygen extraction, was defined as the slope of the StO2 descent to the lowest value. The recovery slope, which is related to microvascular reactivity, was calculated from the deflation of the tourniquet until the recovery of StO2 to the highest value.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged >18 years
* elective on-pump cardiac surgery

Exclusion Criteria:

* pregnancy
* inability to tolerate VOT (e.g., patients with arm deformities, arteriovenous shunts, burns)adult patients aged >18 years scheduled for elective on-pump cardiac surgery
* refusal to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged >18 years scheduled for elective on-pump cardiac surgery in Pusan National University Hospital.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Recovery slope | during applying cardiopulmonary bypass, an average 1-2 hours
  Recovery slope is related to microvascular reactivity, was calculated from the deflation of the tourniquet until the recovery of tissue oxygen saturation to the highest value.
Major adverse events | within postoperative 30 days
  death, acute kidney injury, myocardial infarction, acute respiratory distress syndrome, aggravated heart failure, gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Heon-Jeong Lee, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided